CLINICAL TRIAL: NCT01232270
Title: The Optimal Effect Site Concentration of Propofol for Conscious Sedation in Elderly Male Patients Undergoing Urologic Surgery Under Spinal Anesthesia With or Without Intrathecal Fentanyl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4-2010-0409
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Conscious Sedation Under Spinal Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fentanyl (Active Comparator)
  Interventions: Drug: propofol
- saline (Placebo Comparator)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — 1.1 mcg/ml for initial effect site concentration during spinal anesthesia (The effect site concentration will be changed at each subject by Dixon's up-and-down method.)
  Other Names: Pofol®

SUMMARY:
Since intrathecal fentanyl is known to sedation effect, intrathecal fentanyl will result in lowering propofol requirement for conscious sedation under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* elderly male patients undergoing urologic surgery under spinal anesthesia

Exclusion Criteria:

* patients with any co-morbidity

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Cerebral state index | 1 minute
  every 1 minute(up to 10-minute) after getting effect site concentration of propofol

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Dong Kwon, MD, Ph.D, Principal Investigator — Severance Hospital, Department of Anesthesia and Pain Medicine
Locations (1):
- Severance Hospital, Seoul, South Korea